CLINICAL TRIAL: NCT06115681
Title: Demographic, Clinical Characteristics, and Treatment Outcomes Associated With Dedifferentiated Liposarcoma Patients in China
Brief Title: Real-world Study of Dedifferentiated Liposarcoma Patients in China
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1403-0024
Record Dates: First submitted 2023-10-27; First posted 2023-11-03 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Dedifferentiated Liposarcoma
MeSH Terms: conditions — Liposarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DDLPS patients with 1L treatment at index date (Cohort 1): Patients with unresectable locally advanced or metastatic differentiated liposarcoma (DDLPS) who received at least one line of systemic antineoplastic treatment by the end of cohort identification period (index date = start date of first line (1L) treatment).
- DDLPS patients without 1L treatment at index date (Cohort 2): Patients with DDLPS who have not initiated 1L systemic antineoplastic treatment by the end of cohort identification period (index date = date of initial DDLPS diagnosis during cohort identification period). Patients who initiated 1L treatment afterwards or patients who received adjuvant and/or neoadjuvant therapy only through follow-up were included in Cohort 2.

SUMMARY:
This study will characterize patients with dedifferentiated liposarcoma (DDLPS) in China, including an understanding of demographic, and clinical characteristics as well as treatment patterns and clinical outcomes associated with the current real-world treatment.

ELIGIBILITY:
Inclusion criteria:

* Patient has two or more documented clinical visits in the National Anti-Tumor Drug Surveillance System (NATDSS) network on or after January 1, 2013.
* Patient has a confirmed diagnosis of dedifferentiated liposarcoma (DDLPS) during his/her lifetime.
* At least 18 years old at the date of initial diagnosis.

No exclusion criteria are applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented clinical visits in the National Anti-Tumor Drug Surveillance System (NATDSS) network on or after January 1, 2013 and confirmed dedifferentiated liposarcoma (DDLPS).
Sampling Method: Non-Probability Sample
Enrollment: 1390 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational cohort study conducted to investigate patient characteristics, current treatment patterns and outcomes in Chinese patients with dedifferentiated liposarcoma (DDLPS).
Pre-assignment Details: Only patients diagnosed with DDLPS, who met all the inclusion criteria of having at least 2 documented clinical visits in the National Anti-Tumor Drug Surveillance System (NATDSS) on or after January 1, 2013, and were ≥18 years at initial diagnosis, were included.
Period: Overall Study
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Started | 275 | 1115
Completed | 275 | 1115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients diagnosed with dedifferentiated liposarcoma (DDLPS) who met the inclusion criteria of having at least 2 documented clinical visits in the National Anti-Tumor Drug Surveillance System (NATDSS) in China on or after January 1, 2013 and were aged ≥18 years at initial diagnosis. Eligible patients were identified from January 1, 2013 to December 31, 2021 and were followed from index date until death, end of study period (December 31, 2022), or loss to follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2) | Total
Number analyzed (Participants) | 275 | 1115 | 1390
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (11.5) | 57.4 (11.7) | 57.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 495 | 604
  Male | 166 | 620 | 786
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Secondary Outcome: Cohort 1, Cohort 2: Survival After Initial Diagnosis
Description: Survival after initial diagnosis for each patient was defined as the date of death minus the date of initial diagnosis. For patients with no record of death, survival after initial diagnosis was censored at the last activity date before the end of the study period.
Time Frame: Time from initial diagnosis until the earliest record of death or end of the study period, up to 10 years.
Population: All patients diagnosed with dedifferentiated liposarcoma (DDLPS) who met the inclusion criteria of having at least 2 documented clinical visits in National Anti-Tumor Drug Surveillance System (NATDSS) in China on or after January 1, 2013 and aged ≥18 years at initial diagnosis. Only patients with an existing diagnosis date were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 272 | 1106
months | 30.3 [26.8 to 36.7] | 38.4 [35.0 to 42.6]

2. Secondary Outcome: Cohort 1, Cohort 2: Total Number of Treatment Lines
Description: The total number of treatment lines in both cohorts is reported. Lines of therapy (LOT) were defined by the temporal relationship and sequencing of treatment regimens by using the dates of initiation and discontinuation of chemotherapy, targeted therapy, and/or immunotherapy.
Time Frame: At index date and during follow-up, up to 10 years.
Population: All patients diagnosed with dedifferentiated liposarcoma (DDLPS) who met the inclusion criteria of having at least 2 documented clinical visits in National Anti-Tumor Drug Surveillance System (NATDSS) in China on or after January 1, 2013 and being age ≥18 years at initial diagnosis.
Measure: Median (Inter-Quartile Range); unit: Count of treatment lines per patient
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 275 | 1115
Count of treatment lines per patient | 1.0 [1.0 to 2.0] | 0.0 [0.0 to 0.0]

3. Secondary Outcome: Cohort 1, Cohort 2: First Line (1L) of Therapy by Treatment Type
Description: Number of patients with first line (1L) therapy by treatment type for both cohorts is reported. Lines of therapy (LOT) were defined by the temporal relationship and sequencing of treatment regimens by using the dates of initiation and discontinuation of chemotherapy, targeted therapy, and/or immunotherapy.
Time Frame: At index date and during follow-up, up to 10 years
Population: All patients diagnosed with dedifferentiated liposarcoma (DDLPS) who met the inclusion criteria of having at least 2 documented clinical visits in National Anti-Tumor Drug Surveillance System (NATDSS) in China on or after January 1, 2013 and aged ≥18 years at initial diagnosis. Only patients with non-missing data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 274 | 35
Participants
  Anthracycline-based regimens | 119 | 12
  Anlotinib-based regimens | 85 | 12
  Apatinib-based regimens | 15 | 1
  Immune checkpoint inhibitor only | 10 | 1
  Palbociclib | 9 | 0
  Other | 36 | 9

4. Secondary Outcome: Cohort 1, Cohort 2: Second Line (2L) of Therapy by Treatment Type
Description: Number of patients with second line (2L) therapy by treatment type for both cohorts is reported. Lines of therapy (LOT) were defined by the temporal relationship and sequencing of treatment regimens by using the dates of initiation and discontinuation of chemotherapy, targeted therapy, and/or immunotherapy.
Time Frame: At index date and during follow-up, up to 10 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 114 | 8
Participants
  Anlotinib-based regimens | 37 | 4
  Anthracycline-based regimens | 22 | 2
  Immune checkpoint inhibitor only | 13 | 1
  Apatinib-based regimens | 8 | 0
  Gemcitabine, Docetaxel | 4 | 0
  Other | 30 | 1

5. Secondary Outcome: Cohort 1, Cohort 2: Third Line (3L) of Therapy by Treatment Type
Description: Number of patients with third line (3L) therapy by treatment type for both cohorts is reported. Lines of therapy (LOT) were defined by the temporal relationship and sequencing of treatment regimens by using the dates of initiation and discontinuation of chemotherapy, targeted therapy, and/or immunotherapy.
Time Frame: At index date and during follow-up, up to 10 years
Population: All patients diagnosed with dedifferentiated liposarcoma (DDLPS) who met the inclusion criteria of having at least 2 documented clinical visits in National Anti-Tumor Drug Surveillance System (NATDSS) in China on or after January 1, 2013 and being age ≥18 years at initial diagnosis. Only patients with non-missing data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 51 | 2
Participants
  Anlotinib-based regimens | 16 | 1
  Anthracycline-based regimens | 11 | 1
  Apatinib-based regimens | 5 | 0
  Immune checkpoint inhibitor only | 3 | 0
  Gemcitabine, Docetaxel | 2 | 0
  Other | 14 | 0

6. Secondary Outcome: Cohort 1, Cohort 2: Number of Patients With Treatments Classified as Concurrent Steroid Therapy
Description: Number of patients who received treatments with drugs classified as concurrent steroid therapy for both cohorts is reported.
Time Frame: At index date and during follow-up, up to 10 years
Population: All patients diagnosed with dedifferentiated liposarcoma (DDLPS) who met the inclusion criteria of having at least 2 documented clinical visits in National Anti-Tumor Drug Surveillance System (NATDSS) in China on or after January 1, 2013 and aged ≥18 years at initial diagnosis.
Measure: Count of Participants; unit: Participants
Groups:
- DDLPS Patients Without 1L Treatment at Index Date (Cohort 2): Patients with DDLPS who have not initiated 1L systemic antineoplastic treatment by the end of cohort identification period (index date = date of initial DDLPS diagnosis during cohort identification period). Patients initiated 1L treatment afterwards or patients received adjuvant and/or neoadjuvant therapy only through follow-up will be included in Cohort 2.
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 275 | 1115
Participants | 1 | 1

7. Secondary Outcome: Cohort 1, Cohort 2: Number of Patients With Treatments Classified as Concurrent Immunosuppressant Therapy
Description: Number of patients who received treatments with drugs classified as concurrent immunosuppressant therapy for both cohorts is reported.
Time Frame: At index date and during follow-up, up to 10 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 275 | 1115
Participants | 32 | 2

8. Secondary Outcome: Cohort 1, Cohort 2: Number of Patients With Treatments Classified as Hormone Replacement Therapy
Description: Number of patients who received treatments with drugs classified as hormone replacement therapy for both cohorts is reported.
Time Frame: At index date and during follow-up, up to 10 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
Number analyzed (Participants) | 275 | 1115
Participants | 10 | 0

9. Primary Outcome: Cohort 1: Overall Survival
Description: Overall survival (OS) as an event for each patient in Cohort 1 was defined as the date of death minus the index date or the start day of each line of therapy (LOT). For patients with no record of death, OS was censored at the last activity date before the end of the study period.
Time Frame: Time from index date until the earliest record of death or end of the study period, up to 10 years.
Population: All patients diagnosed with dedifferentiated liposarcoma (DDLPS) who met the inclusion criteria of having at least 2 documented clinical visits in National Anti-Tumor Drug Surveillance System (NATDSS) in China on or after January 1, 2013 and aged ≥18 years at initial diagnosis. Only patients who received at least one line of systemic antineoplastic treatment by the end of cohort identification period were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1)
Number analyzed (Participants) | 275
months
  OS after first line (1L) treatment | 13.4 [12.5 to 15.3]
  OS after second line (2L) treatment: number analyzed (Participants) | 114
  OS after second line (2L) treatment | 11.9 [10.1 to 15.4]
  OS after third line (3L) treatment: number analyzed (Participants) | 51
  OS after third line (3L) treatment | 8.1 [6.0 to 18.2]

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study. All-cause mortality was recorded until end of the observation, up to 10 years.
Description: This was an observational study and was not designed to assess adverse events, therefore safety reporting was not applicable for this study. Adverse events were not planned to be collected as defined in the study protocol. Adverse Events were not monitored/assessed.
Arm/Group | DDLPS Patients With 1L Treatment at Index Date (Cohort 1) | DDLPS Patients Without 1L Treatment at Index Date (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 175/275 | 423/1106
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT06115681/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT06115681/SAP_001.pdf